CLINICAL TRIAL: NCT03916107
Title: Comparison of Different Surgical Treatments for Severe Ptosis Correction RCT Study
Brief Title: Comparison of Different Surgical Treatments for Severe Ptosis Correction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qing-FengLi Li,MD, MD, PhD, Professor, Head of the Department of Plastic and Reconstructive Surgery, Shanghai 9th People'sHospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-81-T72
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Ptosis, Eyelid
Keywords: Ptosis; Frontalis flap
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levator muscle and tarsus resection (Experimental)
  Interventions: Procedure: Levator muscle and tarsus resection
- Frontal muscle flap (Active Comparator)
  Interventions: Procedure: Frontalis flap

INTERVENTIONS:
Procedure: Levator muscle and tarsus resection — Shortening the levator muscle with resection of tarsus to correct severe ptosis
  Arms: Levator muscle and tarsus resection
Procedure: Frontalis flap — Using frontal muscle flap to correct severe ptosis
  Arms: Frontal muscle flap

SUMMARY:
Main research purposes of this research is to compare the therapeutic effect and safety of the superior levator muscle shortening combined with the tarsus resection and the traditional frontal muscle flap in the correction of severe ptosis.

Aside of above we also tend to explore the dose-effect relationship between the amount of levator muscle shortened/ tarsus resection and postoperative ptosis correction amount.So as to develop a more critical and specific guidelines for clinical treatment of ptosis.

So during the research we will recruiting patients with severe ptosis and randomly divide them into levator muscle and tarsus group and frontal muscle flap group, and follow up those patient 6 months post operation so as to evaluate the amount of correction and the side-symptoms.

DETAILED DESCRIPTION:
The ptosis is divided into light, medium and severe according to the difference in muscle strength of the upper levator muscle. According to the previous diagnosis and treatment criteria, for the mild and moderate ptosis, it is recommended to use the method of shortening or partial resection of the levator muscle. For severe patients, because the strength of the upper levator muscles are extremely weak, the function of the upper eye lid can only be reconstructed through the strength of the frontal muscles. So it is recommended to use the frontal muscle flap surgery for correct ptosis. However, compared with the levator levator shortening, the shortcoming of the frontal muscle suspension is to change the nature anatomical relationship of the upper eyelid, resulting in unnatural eye lid lines, obvious frontal lines, easy recurrence and other shortcomings. In the case, this therapy turns out not to be very satisfied.

Based on years of clinical experience in treating ptosis, our research team have tried to use the levator muscle shortening combined with the tarsus resection method for more than 10 years. We have successfully cured more than 1000 patients with severe ptosis and obtained good therapeutic effects. The results are summarized and the sequence is published in several international journals and is recognized by domestic and foreign counterparts. However, for the new procedure of levator muscle shortening combined with tarsus resection, there is currently no comparative study with traditional therapy, and it is impossible to objectively evaluate its efficacy. Secondly, how to improve the long-term effect of levator muscle shortening combined with tarsus resection, whether the eyelid morphology is satisfactory, and the recurrence rate has not been reported. In addition, because the tarsus plays an important role in the shape and function of the eye, including maintaining the function of the tarsus and keeping the cornea moist, etc., the effect of partial removal of the tarsus on the original tarsus function is also worthy of further investigation.

Based on the original clinical results, the project team designed a randomized controlled single-blind study to compare the efficacy and safety of the levator muscle shortening combined with the tarsal resection and the traditional frontal muscle flap in the correction of severe ptosis. At the same time, to explore the dose-effect relationship between the shortening of the levator muscle and the amount of tarsal resection and the amount of correction of the ptosis after operation, the surgical design is more precise and personalized, which provides a scientific basis for further development of clinical diagnosis and treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

* unilateral ptosis patient
* the levator muscle strength less than 4mm
* primary surgery
* older than 3 years
* ocular rectus muscle of good strength;

Exclusion Criteria:

* patients who had undergone ptosis correction surgery
* patients with neurological ptosis, senile ptosis or pseudo ptosis
* patients with abnormal ocular function
* patients with Marcus-Gunn syndromes
* patients with severe systemic disease or intolerant to general anesthesia
* patients or their parents cannot finish follow-up due to educational level or various other reasons.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
levator muscle's strength | 6 months post the treatment
  Measuring the muscle strength: let the patient look straight ahead, the examiner presses the eyebrow arch horizontally with the thumb, interrupting the connection between the frontal muscle and the upper eyelids, and ask patient to look down. Then ask the patient to look up as much as they can, and the scale of this movement is the levator muscle strength.
  When a normal person does not use the frontal muscle, the average scale of the upper eye lids movement is 13.37±2.55mm. The muscle strength of the upper eye lids is generally divided into three levels. The good upper eye lids movement scale is 8mm, the medium is 4~7mm, and the weak one is 0~3mm.
width of eyes | 6 months post the treatment
  Measure the width of eyes while doctor shall make sure patient avoid looking up or using the frontal muscle to lift eyelids.
MRD (margin reflex distance) | 6 months post the treatment
  Measure the distance from the upper temporal margin to the point of reflection at the center of the cornea, while doctor shall make sure patient avoid looking up or using the frontal muscle to lift eyelids.

SECONDARY OUTCOMES:
Numbers of patients not completely corrected | 6 months post the treatment
  Patients who are below:
  1. overcorrection（could result in the inability to close the eye completely）
  2. inadequate correction;
  3. recurrence of ptosis; All above is based on outcome 1,2,3
Numbers of patients having dry eye syndrome | 6 months post the treatment
  using OSDI test to see if patients have dry eye syndrome
Numbers of patients having corneal injury | 6 months post the treatment
  corneal injury using topography to check
Numbers of patients having orbital insufficiency | 6 months post the treatment
  orbital insufficiency, using new national standard visual acuity chart to test
Numbers of patients having conjunctival prolapse; | 6 months post the treatment
  based on examination result using slit-lamp microscope
Numbers of patients having trichiasis; | 6 months post the treatment
  based on examination result using slit-lamp microscope
Numbers of patients having eye infection; | 6 months post the treatment
  based on examination result using slit-lamp microscope

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yang, MD, Phd, Study Director — Shanghai Ninth People's Hospital, Affliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Ninth People's Hospital, Affliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No